CLINICAL TRIAL: NCT02295124
Title: Nausea in Patients Receiving Hydromorphone vs Oxycodone After Total Hip Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0267-AE
Record Dates: First submitted 2013-02-11; First posted 2014-11-20 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Nausea
Keywords: Nausea
MeSH Terms: conditions — Nausea | interventions — Oxycodone; Hydromorphone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone (Active Comparator): Patients will be prescribed oxycodone 10mg (5mg if > age 65) every 2 hours as needed for post-operative pain management in addition to tylenol 1000mg every 6 hours and celecoxib 200mg every 12 hours.
  Interventions: Drug: Oxycodone
- Hydromorphone (Active Comparator): Patients will be prescribed hydromorphone 2mg (1mg if > age 65) every 2 hours as needed in addition to tylenol 1000mg every 6 hours and celecoxib 200mg every 12 hours.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Oxycodone — Patients will receive oxycodone 10mg (5mg if > 65) every 2 hours based on an equianalgesic dose calculation. As per routine practice, the dose will be titrated according to the patient's pain at the discretion of the Acute Pain Service physician who will not be blinded to group allocation.
  Other Names: Supeudol
  Arms: Oxycodone
Drug: Hydromorphone — Patients will receive an initial dose of hydromorphone 2mg (1mg if > 65) every 2 hours as needed based on an equianalgesic dose calculation. As per routine practice, the dose will be titrated according to the patient's pain at the discretion of the Acute Pain Service physician who will not be blinded to group allocation.
  Other Names: Palladone, Dilaudid
  Arms: Hydromorphone

SUMMARY:
The study aims to compare the incidence of side effects caused by Oxycodone and Hydromorphone.

DETAILED DESCRIPTION:
Nausea and vomiting in the post-operative period is considered strongly undesirable by patients and has adverse effects on recovery from outpatient procedures, contributing significantly to delays in discharge from recovery. A know major contributor to the occurrence of post-operative nausea and vomiting is the use of opiate medications which are the cornerstone of post-operative pain management. The investigators hypothesize that the occurrence of this side-effect is different between patients prescribed oxycodone and those receiving hydromorphone for acute pain management after total hip replacement surgery. This investigation is a randomized, double-blind, head-to-head comparison to equipotent administration of oxycodone vs. hydromorphone to determine whether such a difference exists.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification System 1-3
* Age 18-85 years
* Patients undergoing hip replacement surgery under spinal anesthesia

Exclusion Criteria:

* patient refusal
* contraindication or refusal of spinal anesthesia
* inability to provide informed consent
* history of dementia
* intolerance or allergy to oxycodone or hydromorphone
* chronic opioid use or chronic pain disorder
* pregnancy
* history of drug addiction
* history of major psychiatric illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of postoperative nausea | Participants will be followed for the duration of hospital stay, an expected average of 72 hours
  The incidence and severity of nausea will be recorded twice daily up to 72 hours post-operatively

SECONDARY OUTCOMES:
Daily pain scores | 72 hours after surgery
  Pain scores (0-10) will be recorded twice daily until 72 hours post-operatively
Incidence of opioid related itching | 72 hours after surgery
  The presence or absence of the opioid related side effects will be recorded twice daily until 72 hours post-operatively
Incidence of delirium | 72 hours after surgery
  The presence of delirium will be recorded until 72 hours post-operatively
Cumulative in-hospital opioid consumption | 72 hours after surgery
  Total in-hospital opioid consumption in morphine equivalent doses will be calculated for the first 72 hours post-operatively
Use of anti-nausea medications | 72 hours after surgery
  The number of administrations and doses of anti-nausea medications will be evaluated until 72 hours post-operatively
Cumulative drug costs per patient | 72 hours after surgery
  The cumulative drug cost based on all anti-nausea and analgesic medications administered will be calculated for the first 72 hours post-operatively
Post-operative admission duration | Total admission duration, an expected average of 72 hours
  The number of post-operative days required for admission will be assessed. Duration is to be an expected average of 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University of Toronto. University Health Network. Toronto Western Hospital.
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Pavlin DJ, Rapp SE, Polissar NL, Malmgren JA, Koerschgen M, Keyes H. Factors affecting discharge time in adult outpatients. Anesth Analg. 1998 Oct;87(4):816-26. doi: 10.1097/00000539-199810000-00014. PMID 9768776
- [Background] Hartrick C, Van Hove I, Stegmann JU, Oh C, Upmalis D. Efficacy and tolerability of tapentadol immediate release and oxycodone HCl immediate release in patients awaiting primary joint replacement surgery for end-stage joint disease: a 10-day, phase III, randomized, double-blind, active- and placebo-controlled study. Clin Ther. 2009 Feb;31(2):260-71. doi: 10.1016/j.clinthera.2009.02.009. PMID 19302899